CLINICAL TRIAL: NCT00773188
Title: A Single-arm, Open-label, Multicenter Feasibility Trial of Bevacizumab Given in Combination With Concomitant Chemoradiation (Cisplatin and Vinorelbine) in Locally Advanced Unresectable Non-squamous, Non-small Cell Lung Cancer
Brief Title: A Feasibility Trial of Avastin (Bevacizumab) in Combination With Concomitant Chemoradiation (Cisplatin and Vinorelbine) in Patients With Locally Advanced Non-Squamous Non-Small Cell Lung Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO21247
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Bevacizumab; Cisplatin; Vinorelbine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: cisplatin; Drug: vinorelbine

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 7.5mg/kg iv or 15mg/kg iv every 3 weeks
Drug: cisplatin — 75mg/m2 iv according to a standard chemotherapy treatment protocol
Drug: vinorelbine — 15mg/m2 iv according to a standard chemotherapy treatment protocol

SUMMARY:
This single arm study will assess the feasibility of use, safety and tolerability of Avastin(bevacizumab) in combination with chemoradiation therapy in patients with locally advanced unresectable non-squamous non-small cell lung cancer.An initial cohort of patients will receive Avastin 7.5mg/kg iv every 3 weeks, in combination with concurrent thoracic radiation for 6.6 weeks and chemotherapy (cisplatin 75 mg/m2 iv and vinorelbine 15mg/m2 iv administered according to a standard treatment protocol). If no dose-limiting toxicities are observed, a second cohort of patients will receive Avastin at a dose of 15mg/kg iv every 3 weeks, in combination with a similar treatment regimen to that of the first cohort. After 5 cycles of combination treatment, Avastin monotherapy will be administered for a further 4 cycles. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients >=18 years with locoregional advanced unresectable non-squamous NSCLC;
* ECOG performance status of 0 or 1;
* no prior thoracic head and neck irradiation or surgical resection for current lung cancer.

Exclusion Criteria:

* mixed, non-small cell and small cell tumors;
* mixed adeno-squamous carcinomas with a predominant squamous component;
* evidence of tumor invasion or encasement of major vessels;
* history of grade >=2 hemoptysis;
* presence of cavitations in lung lesions at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse events; clinical laboratory parameters; physical exam including vital signs; performance status. | Throughout study

SECONDARY OUTCOMES:
Tumor response | Week 13 and Week 22

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Canada (4):
  - Calgary, Alberta
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario